CLINICAL TRIAL: NCT00208819
Title: Randomized Comparison of Monotherapy (Risperidone, Quetiapine, or Olanzapine) Versus Combination Therapy (Risperidone, Quetiapine, or Olanzapine + Divalproex)in the Management of Dementia With Agitation: A Pilot Comparison of Two Standard Therapies
Brief Title: A Comparison of Two Standard Therapies in the Management of Dementia With Agitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Larry Tune, MD, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0673-2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Senile Dementia, Alzheimer Type; Dementia, Alzheimer Type; Alzheimer Disease; Dementia
Keywords: Alzheimer's Disease; Geriatric; Dementia; Agitation; Behavioral Disturbances; Psychosis
MeSH Terms: conditions — Alzheimer Disease; Dementia; Psychomotor Agitation; Mental Disorders; Psychotic Disorders | interventions — Risperidone; Quetiapine Fumarate; Olanzapine; Valproic Acid

INTERVENTIONS:
Drug: risperidone
Drug: quetiapine
Drug: olanzapine
Drug: divalproex

SUMMARY:
The purpose of this study is to determine whether an antipsychotic medication alone or an antipsychotic medication in combination with divalproex is the most effective and safest way to treat agitation in elderly patients with dementia.

DETAILED DESCRIPTION:
Previous researchers have attempted to establish a "target dose" for antipsychotic medications (such as risperidone, quetiapine, or olanzapine) in treating symptoms of agitation in dementia. They have tried to identify the dose with the best risk-benefit ratio for patients considering the significant side effects the medications can cause. Patients taking the doses identified respond only partially and continue to experience some symptoms of agitation, however. One study showed that in patients whose agitation symptoms were not adequately controlled by the target dose of an antipsychotic medication alone, the addition of divalproex further improved behavior in 72% of patients.

The goal of this study is to compare two standard therapies for the management of agitation symptoms in dementia patients. Subjects in this study will include patients who are admitted to the Wesley Woods Inpatient service for the treatment for dementia complicated by behavioral symptoms. After a patient reaches the target dose of risperidone (up to 1.5 mg/day), quetiapine (up to 175 mg/day), or olanzapine (up to 7.5 mg/day) and agitation symptoms are still not adequately managed, he or she will be randomized to one of two groups. Group 1 participants will continue to receive increasing doses of antipsychotic medication until symptoms are controlled or he or she is unable to tolerate the dose. Group 2 participants will continue to receive the target dose of antipsychotic medication and also receive increasing doses of divalproex until symptoms are controlled or he or she is unable to tolerate the dose. Patients will be evaluated at 4 time points during hospitalization. Patients will be evaluated using scales that measure changes in cognition, function, and behavior. Laboratory and ECG results, and scales testing for movement disorders will be done to monitor safety. The family will then be contacted about 3 months the patient's hospitalization to assess current treatment status, residential status, and health status.

ELIGIBILITY:
Inclusion Criteria:

* inpatients admitted to Wesley Woods Inpatient service for Dementia with psychosis and agitation; taking risperidone (up to 1.5 mg/day), quetiapine (up to 175 mg/day), or olanzapine (up to 7.5 mg/day)

Exclusion Criteria:

* prior sensitivity to risperidone, quetiapine, olanzapine or divalproex

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Agitation Scale (PAS)
DiMarco Rating Scale for Extrapyramidal Symptoms
UKU side effect rating scale:autonomic subscale
Behavioral Activity Rating Scale (BARS)
Visual Analog Scale for Nighttime Sleep and Daytime drowsiness (VAS)
Confusion Assessment Method (CAM)
Mini-Mental State Exam (MMSE)
Cohen-Mansfield Agitation Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Larry E. Tune, MD, MAS, Principal Investigator — Emory University
Locations (1):
- Wesley Woods Geriatric Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Tune L. Management of Noncognitive Symptoms of Dementia. Essentials of Clinical Psychopharmacology, 2nd ed. 2001: 935-948.